CLINICAL TRIAL: NCT01665625
Title: A Prospective Randomized Trial of Regional Versus Systemic Continuous Gemcitabine Chemotherapy in the Treatment of Unresectable Pancreatic Cancer
Brief Title: Regional Versus Systemic Chemotherapy in the Treatment of Unresectable Pancreatic Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Guohong Han, Head of Department of Digestive Interventional Radiology, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XHDD 003
Record Dates: First submitted 2012-07-15; First posted 2012-08-15 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Unresectable Pancreatic Cancer
Keywords: Pancreatic cancer; Intra-arterial infusion; Gemcitabine
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- regional interventional chemotherapy group (Experimental)
  Interventions: Procedure: regional interventional chemotherapy group
- systemic chemotherapy (No Intervention)

INTERVENTIONS:
Procedure: regional interventional chemotherapy group — The patients in experimental group were monitored by X-ray imaging. A 0.038 super-sliding guide wire was inserted after successful puncture, and when site of the pancreatic carcinoma was reconfirmed by conventional angiography, a 5F cobra catheter was used to place the port-catheter drug delivery system in the celiac artery (pancreatic head) or the hepatic artery (pancreatic body and tail). Finally, the port-catheter was embedded under the left upper chest.
  Arms: regional interventional chemotherapy group

SUMMARY:
Systemic chemotherapy with cytotoxic drug is of limited effectiveness in advanced pancreatic cancer patients. Gemcitabine has been used as the first-line drug for advance pancreatic cancer for over two decades and combinations of gemcitabine with different chemotherapeutic drugs have been investigated to improve the outcomes of pancreatic cancer. However, no substantial improvement in patient survival has been achieved. Locoregional chemotherapy via intra-arterial perfusion or chemoemoblization takes advantage of the increasing local drug concentrations and reducing systemic toxicities. In this study, the investigators hypothesis that artery infusion chemotherapy had a better antitumor effect than systemic chemotherapy. The investigators will analyze and evaluate the effect and safety of an implanted percutaneous left subclavian artery port-catheter drug delivery system for regional chemotherapy of inoperable pancreatic carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Karnofsky score > 60,
* Expected survival > 3 months,
* Liver, kidney function and routine blood test within normal range
* No serious cardiopulmonary dysfunction
* No acute infection

Exclusion Criteria:

* Pregnant or lactating women
* Uncontrolled internal diseases
* Past or the presence of other malignancy
* Those who had received immunosuppressive therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2012-08; Primary Completion 2015-08 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
overall surviva | 36 months

SECONDARY OUTCOMES:
Clinical Benefit Rate | 12 months
The median progression-free survival PFS | 12 months
Drug Toxicity | 18 months
  The grading standards of the World Health Organization for acute and subacute toxicity of anticancer drugs will be used to grade toxicity.
surgical complications | 18 months
  Major surgical complications included allergic reaction to the contrast agent, local hematoma, pneumothorax, puncture site bleeding, wound infection, delayed healing or cracking, port-catheter blockage, and necrosis of the tissue surrounding the port-catheter.

CONTACTS AND LOCATIONS:
Overall Officials: Guohong Han, MD, Principal Investigator — Xijing Hospital of Digestive Diseases, Fourth Military Medical University
Locations (1):
- Xijing Hospital of Digestive Diseases, Fourth Military Medical University, Xi'an, Shaanxi, China

REFERENCES:
- [Background] Han GH, Yin ZX, Meng XJ, He CY, Zhang HB, Sun AH, Wu KC, Ding J, Fan DM. Prospective randomized clinical trial of two drug delivery pathway in the treatment of inoperable advanced pancreatic carcinoma. Chin J Dig Dis. 2006;7(1):45-8. doi: 10.1111/j.1443-9573.2006.00243.x. PMID 16412037